CLINICAL TRIAL: NCT03213509
Title: Verbal Autopsy of Maternal Deaths, Stillbirths, and Neonatal Deaths in BetterBirth
Status: Completed | Type: Observational
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Community Empowerment Lab (Other); Population Services International (Other)
Responsible Party: Principal Investigator, Atul Gawande, Principal Investigator, Harvard School of Public Health (HSPH)
Other Study IDs: OPP1017378
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Results first posted 2019-06-05 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Perinatal Death; Neonatal Death; Stillbirth
MeSH Terms: conditions — Perinatal Death; Stillbirth | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Perinatal Death With Pause Point(s) Observed, Intervention Arm: Any perinatal death where one or more pause points was observed by BetterBirth staff (FADA) at 2 months or 6 months post-intervention launch, in the intervention arm of the BetterBirth Trial.
  The study involves administering verbal and social autopsies to the mother or family member of a baby who is in this cohort.
  Interventions: Other: Interview (Social and Verbal Autopsy)
- Perinatal Death With Pause Point(s) Observed, Control Arm: Any perinatal death where one or more pause points was observed by BetterBirth staff (FADA) at 2 months or 6 months post-intervention launch, in the control arm of the BetterBirth Trial.
  The study involves administering verbal and social autopsies to the mother or family member of a baby who is in this cohort.
  Interventions: Other: Interview (Social and Verbal Autopsy)

INTERVENTIONS:
Other: Interview (Social and Verbal Autopsy) — Verbal autopsy is a technique used to determine the cause of death by asking caregivers, friends or family members about signs and symptoms exhibited by the deceased in the period before death. This is usually done using a standardized questionnaire that collects details on signs, symptoms, complaints and any medical history or events. The cause of death, or the sequence of causes that led to death, are assigned based on the data collected by this questionnaire and on any other available information. The social autopsy tool is used in conjunction with the verbal autopsy tool to explore the non-biological factors contributing to a death, including the social, behavioural and health systems determinants of maternal and child deaths.

SUMMARY:
The purpose of this study is to conduct Verbal Autopsies of deaths ( stillbirths and neonatal deaths together) identified in the BetterBirth trial to identify their potential causes, timing, and social determinants.

DETAILED DESCRIPTION:
In order to be included in this study, one must be the mother or family member of an individual who was enrolled in the BetterBirth Trial and died. Women who did not consent to follow-up in the BetterBirth study will be excluded.

We identified these families by using data from the BetterBirth Trial, in which there was a perinatal death where one or more pause points was observed by BetterBirth staff (FADA) at 2 months or 6 months post-intervention launch. Our analyses focus on data surrounding the perinatal deaths.

Respondents for the neonatal deaths and stillbirths include mother or the family members of the baby. Mothers had consented to follow-up as part of the BetterBirth Trial.

These individuals will be initially contacted by telephone. Individuals will be asked to participate in verbal autopsy, and, if they agree, a date and time for the interview will be determined. A data collector from CEL or PSI will visit the participant's home on an agreed-upon date and written consent will be obtained. In the event that participants cannot be reached by phone, study staff members will attempt to make contact via Accredited Social Health Activists (ASHAs), who are appointed by the National Rural Health Mission and act as conduits between patients and the health system. The data collector will attempt to call the relevant ASHA worker and request her assistance in establishing contact with the mother. The ASHA will be asked to provide a telephone number at which the mother can be reached, if possible.

Final attempts at contact will be made via home visit if participants cannot be reached either via telephone or with ASHA engagement. Individuals who are reached at home will be introduced to the study and asked to participate using the appropriate recruitment script. For those individuals who agree to participate, data collectors will schedule a time to return to participants' homes for interviews to be conducted. (Note: Home visits are a culturally acceptable practice in this context; for example, home visits were used in the BetterBirth Trial for collection of 7-day outcomes of mothers and newborns.)

Data will be collected using the WHO standard tools for conducting stillbirth or neonatal verbal autopsies, modified for the local context. A section on social autopsy will also be incorporated in the existing study instrument. These tools are standardized and adapted to use in these settings and have been implemented before in other studies in similar communities in U.P. (example: "AMANHI" and "Impact of topical application of cold-pressed sunflower seed oil with improved massage practices on neonatal mortality: a cluster randomized controlled trial in rural North India"). A team of specially trained data collectors (given the sensitive nature of the verbal autopsy questionnaire) will collect the data on existing Android based data collection platform.

Data will be collected by specially trained data collectors. They will collect the data at participants' homes. Participants will include the mother (in case of neonatal death) and any additional person who was present during the events that led to the death. Additional interviewees may include the delivered mother's husband, mother, mother-in-law, other family member, neighbor, etc. The delivered mother will be asked which individuals, if any, should be included in the interview. The mother and the individuals they indicate will be consented individually but interviewed together.

Each interview will take approximately 60 minutes.

A team of specially trained data collectors will be hired. Data will be collected on tablets using a data collection platform that has in-built checks of missing values, range checks, skip patterns etc. to minimize the error in data collection. A GPS monitoring of location of interview will be conducted. The data will be checked at an aggregate level for heaping, interviewer-specific patterns, etc. Forms identified with errors will be sent back for verification and re-entry, but audit-trail will be captured to ensure that the full trail from original data and changes will be maintained with timestamp, GPS and user information. On-site quality assurance would involve both real-time data checks as well as GPS verification of the location of data collection. Data access will be restricted by users, with different privileges for data collectors, supervisors and study investigators. All personal identification information including names, etc. will be encrypted, and only a unique identification number to identify individuals will be made available for analysis. Data will be hosted over a secured network.

Every case will be coded for assigning underlying cause of death, antecedent causes and timing of death by trained and certified physicians. A WHO standard software and coding protocol will be used by these physicians to assign causes of death. The data collected through tablets will be sent to the central server. The narratives of every case will be collected on paper and a scan of the narrative will be sent along with the data. This entire data will be uploaded on the physician coding software from which the verbal autopsy cases will be allotted to physicians for coding. Each case will be independently coded by two physicians and in case of mismatch in the underlying cause of death between the two physicians, a third physician will independently code for the cause of death. Finally, if none of the three underlying causes of death match, a higher level physician arbitrator will resolve the case - this will be done to minimize unclassified deaths. A physician coordinator, who has extensive prior experience of coding verbal autopsy data will oversee the entire process and resolve issues with the help of supervisors of the data collection team. All the cases will be de-identified before uploading on the software for coding.

The verbal autopsy findings will be helpful to understand the result of the BetterBirth Trial. In addition, the findings will inform future investigations of maternal and newborn harm, especially those further upstream in health system and policy design.

ELIGIBILITY:
Inclusion Criteria:

* Mother, family members, and community members of deceased babies who enrolled in the BetterBirth Trial

Exclusion Criteria:

* Mothers and family members members who did not consent to follow-up in the BetterBirth Trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Respondents for the neonatal deaths and stillbirths include mother, family members, or community members of the baby. Mothers had consented to follow-up as part of the BetterBirth Trial.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2017-08-27 (Actual); Study Completion 2017-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Semrau, PhD, Principal Investigator — Ariadne Labs; Vishwajeet Kumar, Principal Investigator — Community Empowerment Lab; Arti Kumar, Principal Investigator — Community Empowerment Lab; Atul Gawande, MD, MPH, Principal Investigator — Ariadne Labs
Locations (1):
- Community Empowerment Labs, Shivgarh, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: Yes
A de-identified data repository will hold the verbal autopsy data collected, including all data fields collected. At the end of the study, de-identified data will be shared in a public domain.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Please note 170 cases were enrolled (ie, babies who suffered from perinatal mortality). Of these 170 cases, there were four sets of twins, both of whom died. This means that there were a total of 166 potential participants to interview via verbal autopsy (we asked for one interview in the case of twins).
Pre-assignment Details: Note: Perinatal mortality cases were assigned to intervention or control group based on their assignment during the BetterBirth Trial. This assignment did not impact the verbal autopsy data collection process; all cases underwent the same interview process.
Groups:
- Participant Interviewed for Verbal Autopsy, Intervention Arm: Individual who was interviewed about a perinatal death where one or more pause points was observed by BetterBirth staff (FADA) at 2 months or 6 months post-intervention launch, in the intervention arm of the BetterBirth Trial
- Participant Interviewed for Verbal Autopsy, Control Arm: Individual who was interviewed about a perinatal death where one or more pause points was observed by BetterBirth staff (FADA) at 2 months or 6 months post-intervention launch, in the control arm of the BetterBirth Trial
Period: Overall Study
Arm/Group | Participant Interviewed for Verbal Autopsy, Intervention Arm | Participant Interviewed for Verbal Autopsy, Control Arm
Started | 80 | 90
Completed | 76 | 85
Not Completed | 4 | 5
Not completed — Did not consent for verbal autopsy | 4 | 5

BASELINE CHARACTERISTICS:
Population: Participant who consented to be interviewed (verbal autopsy) about a perinatal death where one or more pause points was observed by BetterBirth staff (FADA) at 2 months or 6 months post-intervention launch
Groups:
- Participant Interviewed for Verbal Autopsy, Intervention Arm: Participant interviewed for verbal autopsy regarding a perinatal death where one or more pause points was observed by BetterBirth staff (FADA) at 2 months or 6 months post-intervention launch, in the intervention arm of the BetterBirth Trial
- Participant Interviewed for Verbal Autopsy, Control Arm: Participant interviewed for verbal autopsy regarding a perinatal death where one or more pause points was observed by BetterBirth staff (FADA) at 2 months or 6 months post-intervention launch, in the control arm of the BetterBirth Trial
- Total: Total of all reporting groups
Arm/Group | Participant Interviewed for Verbal Autopsy, Intervention Arm | Participant Interviewed for Verbal Autopsy, Control Arm | Total
Number analyzed (Participants) | 74 | 84 | 158
Age, Categorical [Count of Participants; unit: Participants] — Please note, these age measures refer to the age of the respondent interviewed for the verbal autopsy for each case.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 73 | 84 | 157
    >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 33 [19 to 68] | 31 [18 to 65] | 32 [18 to 68]
Sex: Female, Male [Count of Participants; unit: Participants] — This measure refers to the participants who undertook a verbal autopsy interview.
  Participants
    Female | NA — We did not collect sex of participants who undertook a verbal autopsy interview. | NA — We did not collect sex of participants who undertook a verbal autopsy interview. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Male | NA — We did not collect sex of participants who undertook a verbal autopsy interview. | NA — We did not collect sex of participants who undertook a verbal autopsy interview. | NA — Total not calculated because data are not available (NA) in one or more arms.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  India | 74 | 84 | 158

OUTCOME MEASURES:

1. Primary Outcome: Cause of Death
Description: Cause of perinatal mortality
Time Frame: Early post-natal period (up to 7 days post-partum)
Measure: Count of Participants; unit: Participants
Groups:
- Perinatal Death With Pause Point(s) Observed, Intervention Arm: Any perinatal death where one or more pause points was observed by BetterBirth staff (FADA) at 2 months or 6 months post-intervention launch, in the intervention arm of the BetterBirth Trial
- Perinatal Death With Pause Point(s) Observed, Control Arm: Any perinatal death where one or more pause points was observed by BetterBirth staff (FADA) at 2 months or 6 months post-intervention launch, in the control arm of the BetterBirth Trial
Arm/Group | Perinatal Death With Pause Point(s) Observed, Intervention Arm | Perinatal Death With Pause Point(s) Observed, Control Arm
Number analyzed (Participants) | 76 | 85
Participants
  Stillbirth | 20 | 35
  Early Neonatal Death | 56 | 50

2. Primary Outcome: Cause of Stillbirth
Description: Cause of Stillbirth
Time Frame: Early post-natal period (up to 7 days post-partum)
Measure: Count of Participants; unit: Participants
Arm/Group | Perinatal Death With Pause Point(s) Observed, Intervention Arm | Perinatal Death With Pause Point(s) Observed, Control Arm
Number analyzed (Participants) | 20 | 35
Participants
  Obstructed Labor | 3 | 12
  Other Specific Perinatal Cause | 9 | 9
  Other Obstetric Complication | 2 | 4
  Antepartum Hemorrhage | 3 | 3
  Other | 2 | 3
  Unknown | 1 | 4

3. Primary Outcome: Cause of Early Neonatal Death
Description: Cause of Early Neonatal Death
Time Frame: Early post-natal period (up to 7 days post-partum)
Measure: Count of Participants; unit: Participants
Arm/Group | Perinatal Death With Pause Point(s) Observed, Intervention Arm | Perinatal Death With Pause Point(s) Observed, Control Arm
Number analyzed (Participants) | 56 | 50
Participants
  Perinatal Asphyxia | 26 | 26
  Infection | 13 | 9
  Pre-Term Birth Complications | 8 | 11
  Other Specific Perinatal Cause | 1 | 2
  Congenital Malformations | 3 | 0
  Unknown | 5 | 2

4. Other Pre Specified Outcome: Sex of Babies Who Suffered Perinatal Mortality
Description: This measure refers to the sex of the babies who suffered a perinatal mortality, and whose mother/family member was interviewed about the death via verbal autopsy
Time Frame: Within 7 days postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Perinatal Death With Pause Point(s) Observed, Intervention Arm | Perinatal Death With Pause Point(s) Observed, Control Arm
Number analyzed (Participants) | 76 | 85
Participants
  Male | 41 | 50
  Female | 35 | 35

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the study period (July 3, 2017- August 27, 2017).
Description: There were no adverse events among the individuals who were interviewed for verbal autopsy.
  Please note our outcomes represent cases of perinatal mortality. These cases were expected as our sample was based on perinatal mortality cases from the BetterBirth trial; we performed verbal autopsies on all cases of perinatal mortality in the trial.
Groups:
- Interview (Social and Verbal Autopsy): The study involves administering verbal and social autopsies for BetterBirth Trial Participants who experienced a neonatal or perinatal death.
  Interview (Social and Verbal Autopsy): Verbal autopsy is a technique used to determine the cause of death by asking caregivers, friends or family members about signs and symptoms exhibited by the deceased in the period before death. This is usually done using a standardized questionnaire that collects details on signs, symptoms, complaints and any medical history or events. The cause of death, or the sequence of causes that led to death, are assigned based on the data collected by this questionnaire and on any other available information. The social autopsy tool is used in conjunction with the verbal autopsy tool to explore the non-biological factors contributing to a death, including the social, behavioural and health systems determinants of maternal and child deaths.
Arm/Group | Interview (Social and Verbal Autopsy)
All-Cause Mortality (participants affected / at risk) | 0/170
Serious Adverse Events (participants affected / at risk) | 0/170
Other Adverse Events (participants affected / at risk) | 0/170

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-03-30): https://cdn.clinicaltrials.gov/large-docs/09/NCT03213509/SAP_000.pdf
  • Study Protocol (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/09/NCT03213509/Prot_001.pdf